CLINICAL TRIAL: NCT02266862
Title: Changes in Renal Artery Movement Due to Respiration Before and After Fenestrated Endovascular Repair
Status: Withdrawn | Type: Observational
Why Stopped: No funding
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 14-2330
Record Dates: First submitted 2014-10-13; First posted 2014-10-17 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Fenestrated Endovascular Aortic Repair

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Group: The purpose of this study is to evaluate the location within the renal artery of maximal angular displacement before and after fenestrated endovascular aortic repair (FEVAR) using CT with end-inspiration and end-expiration CT images before and after repair.
  Interventions: Radiation: Study group

INTERVENTIONS:
Radiation: Study group — Patients will receive an additional CT sequence (end-expiration) at the time of their standard CT imaging before and after the repair.

SUMMARY:
Purpose: The purpose of this study is to evaluate the location within the renal artery of maximal angular displacement before and after fenestrated endovascular aortic repair (FEVAR) using CT with end-inspiration and end-expiration CT images before and after repair. Then, the renal artery segment with maximal angular displacement on each will be located and any changes described.

Participants: There will be 30 subjects recruited from UNC Hospitals.

Procedures (methods): For this study, patients will receive an additional CT sequence (end-expiration CT), which will be compared with the standard of care end-inspiration CT to calculate angular displacement and the distance from the aorta.

DETAILED DESCRIPTION:
The investigators would like to evaluate the location within the renal artery of maximal angular displacement before and after fenestrated endovascular aortic repair (FEVAR) using CT with end-inspiration and end-expiration CT images before and after repair. The investigators would then locate the renal artery segment with maximal angular displacement on each and describe any changes. Because these patients would be getting pre and post-surgical CTs as part of standard of care, there would be no added charge to obtain the information for the study. There would be, however, minimal increased radiation exposure resulting from the extra scan being performed during end-expiration and the patients would have to consent to the slight added risk to participate.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing pre-procedural CT scan for FEVAR

Exclusion Criteria:

* Has aortic/renal stent already
* Cannot receive IV contrast due to renal insufficiency or allergy
* Renal arteries are not patent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with fenestrated endovascular aortic repair (FEVAR) will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in angular displacement | Baseline, 6 months
  We will calculate the distance from the aorta and angular displacement both before and after the procedure. Then, a paired t-test will be used to compare these values to determine statistical significance.

CONTACTS AND LOCATIONS:
Overall Officials: Ari Isaacson, MD, Principal Investigator — University of North Carolina, Chapel Hill